CLINICAL TRIAL: NCT07153029
Title: Cognitive Functioning Among Older Adults in Methadone Treatment for Opioid Use Disorder
Brief Title: Older Adults, Methadone, and Cognitive Function
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Bethea A Kleykamp, Assistant Professor, Psychiatry, University of Maryland School of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00116032
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Cognitive Ability General
Keywords: older adults; cognition; feasibility; ecological momentary assessment
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is a prospective feasibility trial evaluating the use of brief, daily, remotely delivered cognitive assessments over 15 consecutive days among patients aged 55 years and older receiving methadone treatment for opioid use disorder (OUD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone-based assessments and cognitive tasks (Experimental): All participants will complete a baseline session to colelct data related to demographics, health history/status, and cognitive functioning. Participants will be oriented to the smartphone application which is delivered via NeuroUX cloud-based technology which send a text message to the smartphone as a prompt for tasks which will be administered across 15 days. All participants complete the same tasks and duration of tasks. Then all participants complete a follow-up assessment to examine their preferences related to the smartphone and cognitive function.
  Interventions: Behavioral: Smartphone based cognitive tasks

INTERVENTIONS:
Behavioral: Smartphone based cognitive tasks — 15 days Smartphone/Cellphone tasks: Using NeuroUX smartphone testing software, Cognitive "games"/tasks lasting approximately 3-4 minutes each will be administered through the a smartphone application and will be prompted via text message twice per day across 15 consecutive days in the morning (8-11am) and evening (5-8). Tasks were chosen to measure aspects of diverse aspects of cognitive that are impaired among patients taking methadone, including N-back task (working memory), the Stroop Task (executive function/cognitive control), and the Variable Difficulty List Memory Test (learning and memory). The 15 days will include two types of task administration: a) Testing Phase: tasks administered at a consistent, fixed difficulty level (days 1-5) b) Remediation Phase: increasing task difficulty in response to participant performance (days 6-15). To encourage adherence, researchers will contact participants to remind them of task completion.

SUMMARY:
The increasing prevalence of opioid use disorder (OUD) among older adults, coupled with high overdose rates and cognitive impairments associated with opioid use, highlights a critical gap in addiction treatment. Cognitive impairments can persist despite treatment and negatively impact recovery outcomes, yet cognitive screening and interventions are rarely integrated into OUD care. This study aims to evaluate the feasibility of remotely delivered, smartphone-based cognitive assessments (administered through NeuroUX web-based software) for older adults (55+) in methadone treatment. The tasks have been "gamified" to make them engaging and brief, which could be appealing to patients. They will complete the tasks for 15 days using the phone provided or their own phone. During days 6-15 of testing, tasks will become incrementally more difficult based on participant performance to assess the feasibility of cognitive training. Cognitive training uses engaging games or tasks to strengthen thinking skills like memory and focus, much like physical exercise strengthens the body. Adherence, acceptability, and usability of the tasks will be assessed. Secondary analyses will explore relationships between task performance and participant characteristics (e.g., baseline cognitive functioning, methadone dose, timing of methadone dose). Findings from this pilot study will provide foundational data for a future grant application to develop and test digital cognitive assessment and training interventions tailored to older adults in addiction treatment. By addressing a critical yet understudied aspect of OUD care this research has the potential to enhance treatment engagement, improve clinical outcomes, and support long-term recovery in the growing older population.

DETAILED DESCRIPTION:
The purpose of this study is to assess cognitive functioning through a smartphone-based application (NeuroUX) across 15 days among patients in methadone treatment for opioid use disorder who are age 55 or older. Aims include:

Aim 1 (Cognitive Testing): For the first 5 days of testing, adherence, acceptability, and useability will be examined after twice daily remote cognitive assessment of executive functioning and learning/memory (N-back, Stroop/Color Trick Task, and Verbal Learning Memory Task) and brief ecological momentary testing (questions that assess recent substance use and craving) among older patients (N=20) in opioid use disorder treatment. Hypothesis: Patients will demonstrate high adherence (> 70% completed assessments), acceptability (> 70% high satisfaction), and usability (mean score > 68 on the "System Usability Scale").

Aim 2 (Cognitive Training): For the days 6-15 of testing, tasks will be made slightly more difficult based on the participants performance (higher performance = more difficulty). Adherence and acceptability (see Aim 1) during this phase of the task and accuracy on tasks will be examined to see if they correspond to number of times completing the task and baseline cognitive assessments. Hypothesis: Patients will demonstrate high adherence and acceptability, and their performance on tasks will increase over time.

Exploratory Aim: examine the relationship between performance on the cognitive tasks and baseline cognitive functioning and follow-up function.

This study is a prospective feasibility trial evaluating the use of brief, daily, remotely delivered cognitive assessments over 15 consecutive days among patients aged 55 years and older receiving methadone treatment for opioid use disorder (OUD). Cognitive assessments will be administered via a study-provided smartphone (or patient's personal phone, depending on preference) using validated tasks targeting executive function (N-back for working memory, Stroop task/Color Trick Task for inhibitory control) and learning/memory (Variable Difficulty List Memory Test). This remote, app-based approach offers a more engaging and less burdensome alternative to traditional, time-intensive in-person cognitive testing commonly used in substance use research. Tasks are designed to be brief (3-4 minutes), visual, engaging, and more aligned with "brain games" than traditional cognitive tasks.

Before starting the daily assessments, participants will attend a baseline session to complete measures of demographics, substance use history and treatment, health characteristics, mood, quality of life, and baseline cognitive performance. During this session, participants will also receive the study smartphone (if they aren't using their own), be oriented to how the tasks will look on their phone, and receive training on completing tasks.

After the 15-day smartphone assessment period, participants will complete a follow-up session that includes repeat measures of mood, quality of life, and cognitive performance, as well as questions about their experience with and perceptions of the smartphone-based cognitive games.

All participants (target number of completers = 20) will complete the same study procedures; no randomization will be used and all study procedures will be transparent to study participants.

ELIGIBILITY:
Inclusion Criteria:

* age 55 and older
* currently in outpatient methadone treatment for opioid use disorder
* participant is alert/able to communicate/able to give acceptable answers on the "Evaluation to Sign Consent form
* participant has normal or correct to normal vision

Exclusion Criteria:

* age 54 or younger
* not in methadone treatment for opioid use disorder

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to smartphone task completion | across 15 days of use
  proportion of completed assessments on the smartphone
Satisfaction with smartphone tasks | across 15 days of use
  Proportion reporting high satisfaction (>70%) with smartphone tasks
Usability of smartphone tasks | after 15 days of use
  mean score > 68 on the "System Usability Scale" a reliable, low-cost usability scale that can be used for global assessments of systems usability. Higher scores indicate greater usability.
Cognitive Task Performance | 15 days of smartphone tasks
  Performance on each of 3 cognitive tasks will be assessed for each time a task is completed. Performance will be compared across days of use.

SECONDARY OUTCOMES:
Laboratory cognitive functioning | 1 month (pre-post 15 day cognitive tasks on smartphone)
  Cognitive functioning in the laboratory before and after smartphone task completion will be assessed using the Iowa Trails Making Task). Changes in performance will be examined pre- and post and analyzed with respect to performance on the smartphone-based cognitive tasks.

OTHER OUTCOMES:
Montreal Cognitive Asesssment (MOCA) (baseline cognitive performance) | Baseline assessment (before 15 days of smartphone task completion)
  The Montreal Cognitive Assessment is a standardized measure of cognitive functioning which will be collected at baseline. We will examine its relationship with smartphone task performance. Higher scores indicate better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- UM Addiction Treatment Programs at 1001 West Pratt, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including baseline characteristics and outcome measures, will be shared with qualified researchers upon request. Data will be available after publication of the primary results. Requests will require approval by the principal investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Start date: date when study is completed and data analyses are completed End date: 5 years from date of study completion and data analyses completed
Access Criteria: Request sent to Principal Investiagator and approved by Principal Investigator